CLINICAL TRIAL: NCT03382652
Title: Continuum™ Metal Bearing System in Total Hip Arthroplasty- A Multi-center, Prospective, Non-controlled Post Market Surveillance Study
Brief Title: Continuum™ Metal Bearing System in Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-H03
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Avascular Necrosis; Osteoarthritis; Inflammatory Arthritis; Post-traumatic; Arthrosis; Total Hip Arthroplasty
Keywords: Total hip arthroplasty; Medical Device; Post Market Surveillance Study; Performance; Safety
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients who received the Continuum Metal on Metal System: Patients requiring total hip arthroplasty, who meet the inclusion/exclusion criteria and received the Continuum Metal on Metal System
  Interventions: Device: Metal-on-Metal Articulation

INTERVENTIONS:
Device: Metal-on-Metal Articulation — <Metal-on-Metal Articulation>: Metasul® Taper Liner and Metasul Femoral Head, <Acetabular Component>:Continuum Acetabular Shell, <Femoral Component>: Zimmer® M/L Taper Hip Stem

SUMMARY:
The study is a multi-center, prospective, non-controlled, consecutive cohort post market surveillance study. The objective of this study is to obtain survival and outcome data on the Continuum Metal Bearing System in primary total hip arthroplasty.

DETAILED DESCRIPTION:
The subject of this clinical investigation is the Continuum Metal Bearing THA System in primary total hip arthroplasty. This system consists of a cementless modular Trabecular Metal® (TM) Continuum Acetabular Shell, a modular Metasul Taper liner, and a modular Metasul femoral head. The characteristics of this THA system may allow for reduction in wear and osteolysis as compared to other approved and marketed THA systems and thus increase the expected implant life.

In total, 3 sites were involved. This number of clinical sites permitted assessment of the consistency among a multitude of investigators. A total number of 83 were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 75 years of age, inclusive.
* Patient is skeletally mature.
* Patient qualifies for primary unilateral or bilateral total hip arthroplasty (THA) based on physical exam and medical history including the following:

  * Avascular necrosis (AVN) Osteoarthritis (OA)
  * Inflammatory arthritis (i.e. Rheumatoid arthritis)
  * Post-traumatic arthritis
* Patient has no history of previous prosthetic replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) of the affected hip joint(s).
* Patient has a Harris Hip Score <70 in the affected hip
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved informed consent.

Exclusion Criteria:

* The patient is:

  * A prisoner
  * Mentally incompetent or unable to understand what participation in the study entails
  * A known alcohol or drug abuser
  * Anticipated to be non-compliant.
* The patient has a neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* The patient has a neurologic condition in the ipsilateral or contralateral limb which affects lower limb function.
* The patient has a diagnosed systemic disease that could affect his/her safety or the study outcome.
* The patient is known to be pregnant.
* The patient is unwilling or unable to give consent, or to comply with the follow-up program.
* The patient has received an investigational drug or device within the previous 6 months.
* The patient has an active or latent infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously. The patient has insufficient bone stock to fix the component. Insufficient bone stock exists in the presence of metabolic bone disease (i.e. osteoporosis), cancer, and radiation. Note: Dual Energy X-ray Absorptiometry (DEXA) may be used to assess the presence of adequate bone stock.
* The patient has known local bone tumors and/or cysts in the operative hip.
* The patient has a known allergic reaction to one or more of the implanted material.
* The patient is Grade III obese with a Body Mass Index (BMI) ≥ 40.
* The patient has osteoradionecrosis in the affected hip joint
* Kidney insufficiency (Kidney insufficiency will be determined based on eGFR value.

See Blood Analysis Report CRF for details)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of max. 100 males and females who require primary total hip arthroplasty. Subjects will be enrolled at 3 investigative centers. Subjects must be geographically accessible throughout the study and be willing and able to attend required follow-up appointments. Candidates who express interest in study participation will be offered informed consent, and eligibility will be determined based upon the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2011-02-09 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (3):
- Saint Davids Medical Center, Austin, Texas, United States
- Finland (2):
  - Jokilaakson terveys oy, Jämsä
  - Hospital District of Southwest Finland, Turku

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Who Received the Continuum Metal on Metal System: Patients requiring total hip arthroplasty, who met the inclusion/exclusion criteria and received the Continuum Metal on Metal System
Period: Overall Study
Arm/Group | Subjects Who Received the Continuum Metal on Metal System
Started | 83
Completed | 44
Not Completed | 39
Not completed — Lost to Follow-up | 6
Not completed — Death | 4
Not completed — Revision | 5
Not completed — Patient withdrew | 3
Not completed — Other reasons | 21

BASELINE CHARACTERISTICS:
Groups:
- Patients Who Received the Continuum Metal on Metal System: Patients required total hip arthroplasty, who met the inclusion/exclusion criteria and received the Continuum Metal on Metal System
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 83
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 57.7 [26.0 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26
  Finland | 57
BMI [Mean (Full Range); unit: kg/m²] | 28.6 [20.3 to 39.8]
Diagnosis [Number; unit: participants]
  Osteoarthritis | 74
  Avascular Necrosis | 7
  Rheumatoid Arthritis | 2

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival at 10 Years
Description: The primary endpoint for this study is implant survival at 10 years which was assessed by revision either of the Continuum Cup or the Metasul liner. A success rate for the experimental group was calculated using the Kaplan-Meier Survival Estimation.
Time Frame: 1, 2, 3, 5, 7, and 10 years postop.
Population: All study patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Patients Who Received the Continuum Metal on Metal System: Patients requiring total hip arthroplasty, who met the inclusion/exclusion criteria and received the Continuum Metal on Metal System
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 83
percentage of participants
  1-year Kaplan Meier Survival Estimate | 98.8 [91.75 to 99.83]
  2-year Kaplan Meier Survival Estimate: number analyzed (Participants) | 79
  2-year Kaplan Meier Survival Estimate | 97.5 [90.34 to 99.37]
  3-year Kaplan Meier Survival Estimate: number analyzed (Participants) | 75
  3-year Kaplan Meier Survival Estimate | 96.16 [88.55 to 98.75]
  5-year Kaplan Meier Survival Estimate: number analyzed (Participants) | 68
  5-year Kaplan Meier Survival Estimate | 96.16 [88.55 to 98.75]
  7-year Kaplan Meier Survival Estimate: number analyzed (Participants) | 56
  7-year Kaplan Meier Survival Estimate | 92.87 [83.58 to 97.00]
  10-year Kaplan Meier Survival Estimate: number analyzed (Participants) | 44
  10-year Kaplan Meier Survival Estimate | 91.01 [80.87 to 95.91]

2. Secondary Outcome: The Harris Hip Score (HHS)
Description: The Harris hip Score (HHS) is an outcome measure that includes a series of questions answered by the patient and physical examinations recorded by a qualified health care Professional. The HHS covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence of deformity (one item, 0-4 points) and range of motion (one item, 0-5 points). The total score can vary from a range of 0 - 100. The outcome score can be categorized as Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70.
Time Frame: Pre-op, 6 weeks, 6 months, 1, 2, 3, 5, 7, and 10 years post-op
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 83
score on a scale
  Preop | 45.1 (12.3)
  6-week: number analyzed (Participants) | 81
  6-week | 85.1 (14.5)
  6-month: number analyzed (Participants) | 77
  6-month | 93.2 (11.3)
  1-year: number analyzed (Participants) | 78
  1-year | 92.2 (12.7)
  2-year: number analyzed (Participants) | 72
  2-year | 93.8 (10.1)
  3-year: number analyzed (Participants) | 71
  3-year | 93.6 (12.9)
  5-year: number analyzed (Participants) | 68
  5-year | 95 (9.0)
  7-year: number analyzed (Participants) | 55
  7-year | 93.5 (11.6)
  10-year: number analyzed (Participants) | 43
  10-year | 91.0 (14.0)

3. Secondary Outcome: The Subject Quality-of-Life (SF-12): Physical and Mental Socres
Description: SF12: The SF-12 is a multipurpose short-form (SF) generic measure of health status. It consists of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). Scores ranges from 0 to 100, with higher scores indicating better physical and mental health functioning.
Time Frame: Pre-op, 6 weeks, 6 months, 1, 2, 3, 5, 7, and 10 years post-op
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 83
score on a scale
  Preop SF-12 (Physical) | 29.8 (7.4)
  6-week SF-12 (Physical): number analyzed (Participants) | 81
  6-week SF-12 (Physical) | 41.8 (8.5)
  6-month SF-12 (Physical): number analyzed (Participants) | 77
  6-month SF-12 (Physical) | 48.4 (9.2)
  1-year SF-12 (Physical): number analyzed (Participants) | 78
  1-year SF-12 (Physical) | 49.5 (9.2)
  2-year SF-12 (Physical): number analyzed (Participants) | 72
  2-year SF-12 (Physical) | 50.0 (8.1)
  3-year SF-12 (Physical): number analyzed (Participants) | 71
  3-year SF-12 (Physical) | 50.7 (8.7)
  5-year SF-12 (Physical): number analyzed (Participants) | 68
  5-year SF-12 (Physical) | 49.5 (9.8)
  7-year SF-12 (Physical): number analyzed (Participants) | 55
  7-year SF-12 (Physical) | 48.8 (10.5)
  10-year SF-12 (Physical): number analyzed (Participants) | 43
  10-year SF-12 (Physical) | 47.9 (9.6)
  Preop SF-12 (Mental) | 52.4 (10.7)
  6-week SF-12 (Mental): number analyzed (Participants) | 81
  6-week SF-12 (Mental) | 56.3 (8.4)
  6-month SF-12 (Mental): number analyzed (Participants) | 77
  6-month SF-12 (Mental) | 56.6 (7.2)
  1-year SF-12 (Mental): number analyzed (Participants) | 78
  1-year SF-12 (Mental) | 56.3 (7.3)
  2-year SF-12 (Mental): number analyzed (Participants) | 72
  2-year SF-12 (Mental) | 57.6 (7.2)
  3-year SF-12 (Mental): number analyzed (Participants) | 71
  3-year SF-12 (Mental) | 57.9 (6.0)
  5-year SF-12 (Mental): number analyzed (Participants) | 68
  5-year SF-12 (Mental) | 57.4 (6.3)
  7-year SF-12 (Mental): number analyzed (Participants) | 55
  7-year SF-12 (Mental) | 55.6 (8.3)
  10-year SF-12 (Mental): number analyzed (Participants) | 43
  10-year SF-12 (Mental) | 57.3 (6.5)

4. Secondary Outcome: Radiographic Evaluations
Description: Radiographic evaluation was performed in order to identify potential adverse events. Investigators at each site were responsible for reviewing the radiological images for any abnormal or significant findings and reporting adverse events if applicable. In addition, an independent radiographic reviewer performed assessments of radiographic films in terms of evidence of radiolucencies, osteolysis, subsidence, acetabular cup migration, and change in acetabular cup angle at 6 months, 1 year and 2 year post-operation. Outcomes included numbers of reported findings per anatomical position and time point.
Time Frame: Immediate-postop, 6 weeks, 6 months, 1, 2, 3, 5, 7, and 10 years post-op.
Population: All study patients
Measure: Number; unit: number of findings
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 83
number of findings
  Total significant findings | 34
  Acetabular side | 6
  Femoral side | 26
  Other | 2
  Immed-postop | 1
  6-week | 5
  6-month | 2
  1-year | 5
  2-year | 6
  3-year | 4
  5-year | 3
  7-year | 6
  10-year | 2

5. Secondary Outcome: Metal Ion Concentration in Blood
Description: Metal ion levels (cobalt, chromium and titanium) were analyzed by an approved Central Laboratory at the time points listed below for all study subjects enrolled in this study. In addition, prior to a revision surgery, a blood draw for metal ion data collection was performed.
Time Frame: Pre-op, 6 months, 1 year, 2 years and 5 years Post-Op.
Population: The numbers of participants listed for metal ion concentrations indicate the number of participants who showed metal ion levels above the detectable limit.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 76
ng/ml
  Preop (Chromium): number analyzed (Participants) | 23
  Preop (Chromium) | 1.1 (0.6)
  6-month (Chromium): number analyzed (Participants) | 52
  6-month (Chromium) | 1.8 (1.0)
  1-year (Chromium): number analyzed (Participants) | 63
  1-year (Chromium) | 2.3 (2.0)
  2-year (Chromium): number analyzed (Participants) | 59
  2-year (Chromium) | 2.4 (1.6)
  5-year (Chromium): number analyzed (Participants) | 61
  5-year (Chromium) | 2.2 (1.3)
  Preop (Cobalt): number analyzed (Participants) | 19
  Preop (Cobalt) | 1.2 (1.1)
  6-Month (Cobalt): number analyzed (Participants) | 31
  6-Month (Cobalt) | 2.2 (1.4)
  1-year (Cobalt): number analyzed (Participants) | 38
  1-year (Cobalt) | 2.9 (3.6)
  2-year (Cobalt): number analyzed (Participants) | 38
  2-year (Cobalt) | 2.2 (1.1)
  5-year (Cobalt): number analyzed (Participants) | 38
  5-year (Cobalt) | 2.3 (1.9)
  Preop (Titanium): number analyzed (Participants) | 21
  Preop (Titanium) | 4.9 (1.2)
  6-month (Titanium): number analyzed (Participants) | 21
  6-month (Titanium) | 5.4 (1.9)
  1-year (Titanium): number analyzed (Participants) | 3
  1-year (Titanium) | 6.1 (0.7)
  2-year (Titanium): number analyzed (Participants) | 6
  2-year (Titanium) | 4.6 (2.3)
  5-year (Titanium): number analyzed (Participants) | 66
  5-year (Titanium) | NA (0) — At 5 years post-surgery all patients had titanium ion concentrations below the detectable limit of <5.0 ng/ml.

6. Secondary Outcome: EQ5D
Description: EQ5D: The EQ-5D is a standardized Instrument widely used to measure health status. It is a self reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes 5 questions referring to mobility, self care, daily activities, pain/discomfort, and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. In the derived EQ-5D-5L score, the highest score is 1 and the lowest score is -0.573; negative numbers correspond to a self-assessed health state worse than being dead. The VAS is a vertical scale ranging from 100 ('The best health you can imagine') to 0 ('The warst health you can imagine') where the patient reports his/her self-rated health.
Time Frame: Pre-op, 6 weeks, 6 months, 1, 2, 3, 5, 7, and 10 years post-op
Population: All study patients. At preoperative, EQ-5D scores of only 57 patients (not collected at the US site) were available for this report.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 57
units on a scale
  Preop EQ-5D-5L | 0.6 (0.2)
  6-week EQ-5D-5L | 0.8 (0.1)
  6-month EQ-5D-5L: number analyzed (Participants) | 56
  6-month EQ-5D-5L | 0.9 (0.1)
  1-year EQ-5D-5L: number analyzed (Participants) | 55
  1-year EQ-5D-5L | 0.9 (0.1)
  2-year EQ-5D-5L: number analyzed (Participants) | 55
  2-year EQ-5D-5L | 1.0 (0.1)
  3-year EQ-5D-5L: number analyzed (Participants) | 54
  3-year EQ-5D-5L | 1.0 (0.1)
  5-year EQ-5D-5L: number analyzed (Participants) | 49
  5-year EQ-5D-5L | 0.9 (0.2)
  7-year EQ-5D-5L: number analyzed (Participants) | 47
  7-year EQ-5D-5L | 0.9 (0.1)
  10-year EQ-5D-5L: number analyzed (Participants) | 43
  10-year EQ-5D-5L | 0.9 (0.2)

7. Secondary Outcome: Creatine Concentration and BUN
Description: Renal function (BUN and Creatinine) were analyzed by an approved Central Laboratory at the time points listed below for all study subjects enrolled in this study. In addition, prior to a revision surgery, a blood draw for metal ion data collection was performed.
Time Frame: Pre-op, 6 months, 1 year, 2 years and 5 years Post-Op.
Population: The numbers of participants listed for renal function demonstrated the number of participants tested.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 76
mg/dl
  Preop (Creatine): number analyzed (Participants) | 75
  Preop (Creatine) | 0.8 (0.2)
  6-month (Creatine): number analyzed (Participants) | 74
  6-month (Creatine) | 0.8 (0.2)
  1-year (Creatine) | 0.9 (0.2)
  2-year (Creatine): number analyzed (Participants) | 65
  2-year (Creatine) | 0.9 (0.2)
  5-year (Creatine): number analyzed (Participants) | 65
  5-year (Creatine) | 0.9 (0.2)
  Preop (BUN): number analyzed (Participants) | 70
  Preop (BUN) | 14.9 (4.9)
  6-month (BUN): number analyzed (Participants) | 72
  6-month (BUN) | 14.3 (5.1)
  1-year (BUN) | 14.1 (5.0)
  2-year (BUN): number analyzed (Participants) | 65
  2-year (BUN) | 14.2 (5.9)
  5-year (BUN): number analyzed (Participants) | 61
  5-year (BUN) | 15.2 (4.5)

8. Secondary Outcome: Calculated GFR
Description: Renal function (BUN, Creatinine and GFR) were analyzed by an approved Central Laboratory at the time points listed below for all study subjects enrolled in this study. In addition, prior to a revision surgery, a blood draw for metal ion data collection was performed.
Time Frame: Pre-op, 6 months, 1 year, 2 years and 5 years Post-Op.
Population: The numbers of participants listed for renal function demonstrated the number of participants tested.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²
Arm/Group | Patients Who Received the Continuum Metal on Metal System
Number analyzed (Participants) | 76
mL/min/1.73 m²
  Preop (GRF): number analyzed (Participants) | 74
  Preop (GRF) | 99.3 (34.5)
  6-month (GRF): number analyzed (Participants) | 74
  6-month (GRF) | 101.8 (26.4)
  1-year (GRF) | 98 (23.8)
  2-year (GRF): number analyzed (Participants) | 65
  2-year (GRF) | 92.1 (24.0)
  5-year (GRF): number analyzed (Participants) | 65
  5-year (GRF) | 83.4 (16.0)

ADVERSE EVENTS:
Time Frame: Safety was evaluated by monitoring the frequency and incidence of adverse events (AE), serious adverse events (SAE), adverse device effects (ADE) and serious adverse device effects (SADE) throughout the participation of the study from enrollment to 10-year follow-up
Description: Adverse Events and Adverse Device Effects were documented during the whole course of the study.
Arm/Group | Patients Who Received the Continuum Metal on Metal System
All-Cause Mortality (participants affected / at risk) | 4/83
Serious Adverse Events (participants affected / at risk) | 25/83
Other Adverse Events (participants affected / at risk) | 62/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received the Continuum Metal on Metal System (N=83)
Other General Complication (General disorders) | 7 (7)
Oncological events (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Neurological events (Nervous system disorders) | 3 (3)
Cardiovascular events (Cardiac disorders) | 5 (5)
Musculoskeletal (non-hip) events (Musculoskeletal and connective tissue disorders) | 4 (6)
Dermatological events (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary/Respiratory events (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (hip), superficial (Infections and infestations) | 1 (1)
Gastrointestinal events (Gastrointestinal disorders) | 1 (1)
Delayed Wound Healing (Surgical and medical procedures) | 1 (1)
Instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Endocrine (Endocrine disorders) | 1 (1)
Infection (non-hip) (Infections and infestations) | 1 (1)
ENT (Ear and labyrinth disorders) | 1 (1)
Dislocation (Musculoskeletal and connective tissue disorders) | 1 (1)
Other Hip Related Radiographic Finding (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received the Continuum Metal on Metal System (N=83)
Musculoskeletal (non-hip) (Musculoskeletal and connective tissue disorders) | 35 (58)
Other General Complication (General disorders) | 15 (19)
Thigh/Groin/Hip Pain (Musculoskeletal and connective tissue disorders) | 15 (22)
Cardiovascular (Cardiac disorders) | 10 (13)
Gastrointestinal (Gastrointestinal disorders) | 9 (11)
Genitourinary / Renal (Renal and urinary disorders) | 7 (7)
Other Hip Related Radiographic Finding (Musculoskeletal and connective tissue disorders) | 7 (7)
Neurological (Nervous system disorders) | 5 (7)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dermatological (Skin and subcutaneous tissue disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
The US site was terminated after the 7-year follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT03382652/Prot_SAP_000.pdf